CLINICAL TRIAL: NCT03814226
Title: The Effect of PACAP-38 Infusion in Inducing Headache in Patients With Cluster Headache
Brief Title: PACAP-38 Infusion in Patients With Cluster Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Agneta Snoer, MD, PhD Student, Investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-17011569
Record Dates: First submitted 2019-01-15; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACAP-38 infusion (Experimental): According to main hypothesis PACAP-38 is expected to induce headache. PACAP-38 causes marked vasodilation visible to investigator. PACAP38 (10 pmol/kg/min) is infused over 20 minutes, patients are observed before (15 minutes), during and after (70 minutes) infusion. Blood samples are drawn at fixed time-points.
  Interventions: Other: Evaluation of headache inducing capabilities of PACAP38
- VIP infusion (Active Comparator): According to main hypothesis VIP is not expected to induce headache. VIP also causes marked vasodilation visible to investigator, which is why VIP is chosen as an active comparator. VIP (10 pmol/kg/min) is infused over 20 minutes. VIP is infused over 20 minutes, patients are observed before (15 minutes), during and after (70 minutes) infusion. Blood samples are drawn at fixed time-points.
  Interventions: Other: Evaluation of headache inducing capabilities of PACAP38

INTERVENTIONS:
Other: Evaluation of headache inducing capabilities of PACAP38 — We wish to investigate the headache inducing capabilities of PACAP-38, a vasoactive peptide, over a 20 minute infusion. As PACAP-38 casues visible vasodilation, another vasoactive peptide, called VIP will be used as an active comparator.

SUMMARY:
A randomized, double-blinded, two-way crossover study investigating the headache inducing capabilities of PACAP-38 in patients with cluster headache. Forty-five patients (15 episodic patients in cluster, 15, episodic patients in remission and 15 chronic cluster headache patients) are expected to participate. Each patients will on two separate study days in a randomized way receive an infusion of PACAP-38 and VIP over 20 minutes followed by an observation period of 70 minutes. Blood samples for investigation of VIP, PACAP38; CGRP, NSE, Histamine and Tryptase will be drawn at fixed time-points during experiment.

ELIGIBILITY:
Inclusion Criteria:

* Episodic or chronic cluster headache according to international classification of headache disorders
* Age 18-65 years
* Weight 50-100 kg
* If women of childbearing potential, then must use safe contraceptives

Exclusion Criteria:

* Episodic tension-type headache > 15 days per month
* Other primary headache disorders, except tension-type headache < 5 days per month
* Episodic cluster headache patients outside cluster must be completely headache free a minimum of 8 hours prior to experiment
* Episodic cluster headache patients in cluster and chronic cluster headache patients must be completely headache free a minimum of 4 hours prior to experiment
* Current or recent use (30 days) of injected or oral corticosteroids
* Pregnant or lactating women
* A history or clinical signs of hypertension (BP > 150mmHg systolic / 100mmHg diastolic)
* A history or clinical signs of hypotension (BP <90 mmHg systolic / 50mmHg diastolic)
* A history of cardiovascular or cerebrovascular disease
* A history of psychiatric disease or substance abuse
* A medical history or clinical signs of disease that according to investigator would preclude participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-05-05 (Estimated)

PRIMARY OUTCOMES:
Headache | 90 minutes
  Difference in incidence of headache within 90 minutes of infusion between PACAP-38 infusion and VIP infusion
Plasma/serum levels of PACAP-38, VIP, CGRP, Histamine, Tryptase and NSE | 90 minutes
  Changes in plasma/serum concentrations of the following markers after infusion of PACAP-38 and VIP: PACAP-38, VIP, CGRP, Histamine, Tryptase, NSE
Plasma/serum levels of PACAP-38, VIP, CGRP, Histamine, Tryptase and NSE after infusion | 90 minutes
  Difference in plasma/serum concentrations of the following markers after infusion of PACAP-38 and VIP: PACAP-38, VIP, CGRP, Histamine, Tryptase, NSE between patients with induced cluster headache and patients without headache
Plasma/serum levels of PACAP-38, VIP, CGRP, Histamine, Tryptase and NSE at baseline | 90 minutes
  Difference in plasma/serum concentrations of the following markers at baseline: PACAP-38, VIP, CGRP, Histamine, Tryptase, NSE between patients with episodic cluster headache in remission, episodic cluster headache in cluster, and chronic cluster headache
Headache intensity | 90 minutes
  Difference in AUD for headache intensity scores (0-90 minutes)
Time to headache peak | 90 minutes
  Difference in time to peak headache between PACAP-38 day and VIP day

SECONDARY OUTCOMES:
Change in mean arterial blood pressure | 90 minutes
  Difference in area under the curve (AUC) for mean arterial pressure (based on systolic and diastolic measurements) and heart rate during experiment
Plasma/serum levels of PACAP-38, VIP, CGRP, Histamine, Tryptase and NSE | Baseline
  Difference in serum/plasma levels of PACAP-38, VIP, CGRP, Histamine, Tryptase and NSE at baseline in patients who develop a cluster headache attack compared to those who do not

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, Professor, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Deligianni C, Pellesi L, Chaudhry BA, Haulund Vollesen AL, Snoer AH, Hannibal J, Jensen RH, Ashina M. Plasma levels of VIP are not elevated during PACAP- and VIP-induced cluster headache attacks: an exploratory study. Front Neurol. 2023 Apr 18;14:1135246. doi: 10.3389/fneur.2023.1135246. eCollection 2023. PMID 37143998
- [Derived] Pellesi L, Chaudhry BA, Vollesen ALH, Snoer AH, Baumann K, Skov PS, Jensen RH, Ashina M. PACAP38- and VIP-induced cluster headache attacks are not associated with changes of plasma CGRP or markers of mast cell activation. Cephalalgia. 2022 Jul;42(8):687-695. doi: 10.1177/03331024211056248. Epub 2021 Nov 25. PMID 34822741
- [Derived] Vollesen ALH, Snoer A, Chaudhry B, Petersen AS, Hagedorn A, Hoffmann J, Jensen RH, Ashina M. The effect of pituitary adenylate cyclase-activating peptide-38 and vasoactive intestinal peptide in cluster headache. Cephalalgia. 2020 Nov;40(13):1474-1488. doi: 10.1177/0333102420940689. Epub 2020 Sep 22. PMID 32962406